CLINICAL TRIAL: NCT04013815
Title: Erector Spinae Plane Block Versus Intrapleural Intercostal Plane Block for Post-thoracotomy Pain: a Randomized Trial
Brief Title: Erector Spinae Plane Block for Post-thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Silvia Fiorelli, principal investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESP
Record Dates: First submitted 2019-07-03; First posted 2019-07-10 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Pain, Postoperative
Keywords: erector spinae plane block; thoracotomy; ultrasound guided nerve block; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: 60 patients will be enrolled to undergo thoracotomy lung resection surgery.
  The population will be divided into two groups based on the type of block made:
  Group E: ESP block (n = 30)
  Group I: Intercostal block (n = 30)
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and investigator checking the pain are not aware of which block has been performed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group E (Experimental): patients receiving the ESP block
  Interventions: Procedure: erector spinae plane block with ropivacaine
- group I (Active Comparator): patients receiving the intercostal nerve block
  Interventions: Procedure: Intercostal nerve block with ropivacaine

INTERVENTIONS:
Procedure: erector spinae plane block with ropivacaine — The block is performed immediately before surgery. by an ultrasound guide, with the probe positioned longitudinally, the spinous process of T5 is identified. A peripheral block needle is inserted in the cephalo-caudal direction (caliber 21G and length 10 cm) and 3 ml of physiological solution are injected to confirm the injection site: fascial plane between the erector spinae muscle and the large rhomboid, near the tip of the transverse process of T5. Once the correct position of the needle tip has been confirmed, ropivacaine 0.75% 20 ml is injected.
  Arms: group E
Procedure: Intercostal nerve block with ropivacaine — The intercostal nerve block will be performed by the surgeon at the time of thoracotomy from the 4th to the 8th intercostal space, by injecting 20 ml of 0.75% ropivacaine (4 ml for each space). The injection is performed at about 2-3 cm from the spine.
  Arms: group I

SUMMARY:
Post-thoracotomy pain is one of the most severe forms of post-operative pain. Among the most common techniques for the management of post-thoracotomy pain, there are the intercostal nerve block, and a recently described block, the erector spinae plane block (ESP).To date, there are no studies that compare the efficacy of ESP block with other pain relief methods in acute post-thoracotomy pain. The objective of this randomized study is to compare the analgesic efficacy of these two techniques in the control of acute post-thoracotomy chest pain, block of erector spinae vs intrapleural intercostal block.

DETAILED DESCRIPTION:
Post-thoracotomy pain is one of the most severe forms of post-operative pain that can be attributed to muscle incision, rib retraction or resection, and damage to the intercostal nerves. Inadequate control of this post-operative pain can contribute to a deterioration of the respiratory function, with limitation of the ventilation, appearance of atelectasis, ineffective cough, and increased risk of infectious complications. Moreover, recent evidence shows that persistent pain after surgery, in addition to being responsible for chronic post-surgical pain syndrome, is associated with a delay in post-operative recovery and a return to normal daily life activities. The most common techniques for the management of post-thoracotomy pain are in addition to systemic intravenous analgesia, thoracic epidural, paravertebral nerve block and intercostal nerve block. Although the thoracic epidural has been considered for years the gold standard for the control of post-operative pain following thoracotomy, it is not risk-free, requires an expert operator, and can be contraindicated in some categories of patients. The intercostal nerve block, performed through the injection of the local anesthetic in multiple intercostal spaces before performing thoracotomy, may be one of the alternatives to a thoracic epidural in terms of safety and efficacy and is technically easy and quick to perform. This block is found to be particularly effective in reducing post-operative pain when associated with a mini-thoracotomy, helping to improve the outcome of patients undergoing major lung resection. A technique of more recent description (2016) is the erector spinae plane block (ESP) . This interfascial block is performed in the posterior thoracic region homolaterally at the site of the intervention at the level of the T5 transverse process (fifth thoracic vertebra), the ultrasound marker of the block. The ESP block is easy and safe to perform thanks to the ultrasound-guided method and the absence of vascular-nerve structures at risk of damage in the vicinity of the injection site and allows analgesia of the posterior and anterolateral thoracic wall and of the axillary region. In fact, cadaveric studies have shown an anesthetic distribution both in the cranial caudal sense (T2-T8) along the fascia between erector spinae and large rhomboid, and in the anteroposterior direction, with the blockage of the spinal thoracic nerve roots. ESP block was described in the treatment of chronic chest pain in the first place, but was subsequently used as rescue therapy in acute post-thoracotomy pain; it has also been tested in upper abdominal surgery, performed bilaterally. Use in four cases of acute post video thoracoscopy pain management has also been described. Recently, some randomized controlled trials have been carried out that showed: greater analgesic efficacy of ESP compared to intravenous multimodal analgesia standard for the treatment of post-operative pain, with less recourse to rescue doses of morphine following laparoscopic cholecystectomy, mastectomy and cardiac surgery. To date, there are no studies that compare its efficacy with other pain relief methods in acute post-thoracotomy pain. The objective of our study is to compare the analgesic efficacy of these two techniques in the control of acute post-thoracotomy chest pain, blockade of erector spinae vs intrapleural intercostal blockade.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracotomy lung resection surgery between 45 and 80 years

Exclusion Criteria:

* Patients allergic to the drugs used in the study
* Patients with diabetic neuropathy
* Patients with severe hepatic or renal insufficiency
* emergent surgery
* Age <45 years or> 80 years

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 12 hours from surgery
  efficacy measured through the evaluation of the NRS score (Numerical Rating Scale) , that ranges from '0' representing one pain extreme (e.g. " no pain") to '10' representing the other pain extreme

SECONDARY OUTCOMES:
opioid consumption | through surgery completed
  the amount of opioid used during the surgical procedure (remifentanil, mcg)
function and strength of the respiratory muscle | 12 hours from the surgery
  respiratory pressure meter measuring MIP (maximal inspiratory pressure) and MEP (maximal expiratory pressure)
patient satisfaction about the analgesia technique | 12 hours after surgery
  Likert satisfaction scale,Satisfaction rate ranged from 5 meaning highly satisfied to 1 meaning highly unsatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Sant Andrea Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Loan WB, Morrison JD. The incidence and severity of postoperative pain. Br J Anaesth. 1967 Sep;39(9):695-8. doi: 10.1093/bja/39.9.695. No abstract available. PMID 6051231
- [Background] Sabanathan S, Eng J, Mearns AJ. Alterations in respiratory mechanics following thoracotomy. J R Coll Surg Edinb. 1990 Jun;35(3):144-50. PMID 2203902
- [Background] Nunn JF. Effects of anaesthesia on respiration. Br J Anaesth. 1990 Jul;65(1):54-62. doi: 10.1093/bja/65.1.54. No abstract available. PMID 2200485
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Sabanathan S, Smith PJ, Pradhan GN, Hashimi H, Eng JB, Mearns AJ. Continuous intercostal nerve block for pain relief after thoracotomy. Ann Thorac Surg. 1988 Oct;46(4):425-6. doi: 10.1016/s0003-4975(10)64657-7. PMID 3178353
- [Background] D'Andrilli A, Ibrahim M, Ciccone AM, Venuta F, De Giacomo T, Massullo D, Pinto G, Rendina EA. Intrapleural intercostal nerve block associated with mini-thoracotomy improves pain control after major lung resection. Eur J Cardiothorac Surg. 2006 May;29(5):790-4. doi: 10.1016/j.ejcts.2006.01.002. Epub 2006 Feb 14. PMID 16481188
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152
- [Background] Luis-Navarro JC, Seda-Guzman M, Luis-Moreno C, Lopez-Romero JL. The erector spinae plane block in 4 cases of video-assisted thoracic surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Apr;65(4):204-208. doi: 10.1016/j.redar.2017.12.004. Epub 2018 Jan 11. English, Spanish. PMID 29336785
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Background] Krishna SN, Chauhan S, Bhoi D, Kaushal B, Hasija S, Sangdup T, Bisoi AK. Bilateral Erector Spinae Plane Block for Acute Post-Surgical Pain in Adult Cardiac Surgical Patients: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):368-375. doi: 10.1053/j.jvca.2018.05.050. Epub 2018 Jun 4. PMID 30055991